CLINICAL TRIAL: NCT01631136
Title: Phase III Study Evaluating Two Strategies of Maintenance, One With Pemetrexed in Continuous Strategy and One According to the Response of Induction Chemotherapy, in Non Squamous Non Small Cell Lung Cancer of Advanced Stage
Brief Title: Strategies for Maintenance Therapies in Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-GFPC-1101
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; IFCT; Maintenance; Switch
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous maintenance Therapy (Active Comparator): Induction chemotherapy by cisplatin + pemetrexed and maintenance therapy by pemetrexed
  Interventions: Drug: Cisplatin; Drug: Pemetrexed
- Maintenance according to the response of induction (Experimental): Induction chemotherapy by cisplatin + gemcitabine followed by :
  * continuous maintenance therapy by gemcitabine if response disease
  * switch maintenance therapy by pemetrexed if stable disease
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Cisplatin — 75 mg/m²
  Arms: Continuous maintenance Therapy
Drug: Pemetrexed — 500 mg/m²
Drug: Cisplatin — 80 mg/m²
  Arms: Maintenance according to the response of induction
Drug: Gemcitabine — 1250 mg/m²
  Arms: Maintenance according to the response of induction

SUMMARY:
In France, lung cancer is responsible for more than 30000 each year. Progress was made in treatment of lung cancer in the last five years due to targeted therapies and to strategical evolutions consisting in a best adjustment of treatments. Maintenance strategies is one of this strategical evolution. It is based on maintaining continuous therapeutical pression in order to preserve the therapeutical benefit obtained by the first line (induction chemotherapy). Several clinical trials showed that maintenance strategies increase the duration of controlled disease.

There is two types of maintenance strategies:

* Continuous maintenance : prolongation of the treatment initially associated with platin until progression
* Switch maintenance : introduction of a new treatment after the end of induction chemotherapy

The aim of this study is to compare two maintenance strategies

* A continuous maintenance by pemetrexed
* A switch maintenance or a continuous maintenance according to the response of induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-squamous NSCLC histologically or cytologically confirmed
* Stage IV with a cytologically or histologically confirmation for an unique metastasis
* No EGFR activating mutation or indeterminate EGFR mutational status
* At least one measurable lesion
* Age between 18 and 70
* PS 0 or 1

Exclusion Criteria:

* squamous cell lung cancer, small cell lung cancer , neuroendocrine cell lung cancer
* Knowledge of ALK gene rearrangement
* Symptomatic central nervous system metastases or requiring immediate cerebral radiotherapy
* Superior venous cave syndrome except if treated by implantation of a prosthesis
* Previous anti-tumoral treatment
* Concomitant radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 932 (Actual)
Dates: Start 2012-07; Primary Completion 2017-05-02 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | around 20 months

SECONDARY OUTCOMES:
Disease free survival | Around 5 months
Control and response rate | After 4 cycles
Safety analysis | Around 5 months
  Number of patients with at least one adverse event in each arm and number of adverse events with the relationship, intensity and the cycle of appearance
treatment exposure | Around 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Maurice PEROL, MD, Principal Investigator — Centre Léon Bérard, Lyon; Pierre-Jean SOUQUET, MD, PhD, Principal Investigator — Centre Hospitalier Lyon Sud
Locations (91):
- France (91):
  - Abbeville - CH, Abbeville
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Clinique Claude Bernard, Albi
  - Annemasse - CH, Ambilly
  - Angers - CHU, Angers
  - Annecy - CH, Annecy
  - Hôpital Privé d'Antony, Antony
  - Argenteuil -CH, Argenteuil
  - Aubenas - CH, Aubenas
  - CH de la Côte Basque, Bayonne
  - Beauvais - CH, Beauvais
  - CHU Besancon - Pneumologie, Besançon
  - Béziers - CH, Béziers
  - Hôpital Ambroise Paré - Pneumologie, Boulogne
  - Caen - Centre François Baclesse, Caen
  - Caen - CHU Côte de Nacre, Caen
  - Cahors - CH, Cahors
  - CH de Cannes, Cannes
  - Castelnau Le Lez - Clinique, Castelnau
  - CH Chambery, Chambéry
  - Charleville-Mézières - CH, Charleville-Mézières
  - Centre Hospitalier, Chauny
  - CH, Cholet
  - Hôpital Percy-Armées - Pneumologie, Clamart
  - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Creil - GHPSO, Creil
  - CHI Créteil, Créteil
  - CH de Dax, Dax
  - Centre d'Oncologie du Parc, Dijon
  - Centre Georges François Leclerc, Dijon
  - Draguignan - CH, Draguignan
  - Grenoble - CHU, Grenoble
  - Saint Omer - CHI, Helfaut
  - CH de Jonzac, Jonzac
  - La Roche Sur Yon - CH, La Roche-sur-Yon
  - Le Mans - Centre Hospitalier, Le Mans
  - CHU (Hôpital Calmette) - Pneumologie, Lille
  - Lille - GHPSO, Lille
  - Limoges - Hôpital du Cluzeau, Limoges
  - CH de Longjumeau, Longjumeau
  - Centre Léon Bérard, Lyon
  - CH Saint Joseph Saint Luc, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Louis Pradel, Lyon
  - Lyon - Hôpital Jean Mermoz, Lyon
  - Hôpital Nord - Oncologie Multidisciplinaire & Innovations Thérapeutiques, Marseille
  - Maubeuge - Polyclinique du Parc, Maubeuge
  - CH de Macon, Mâcon
  - Meaux - CH, Meaux
  - Mont de Marsan - CH, Mont-de-Marsan
  - Centre Hospitalier, Montélimar
  - Montpellier - Clinique Clémentville, Montpellier
  - Mulhouse - CH, Mulhouse
  - Nancy - polyclinique Gentilly, Nancy
  - CHU Nancy, Nancy
  - Nevers - CH, Nevers
  - Nice - CAC, Nice
  - Orléans - CH, Orléans
  - Paris - Saint Louis, Paris
  - Hopital Tenon - Pneumologie, Paris
  - GH Paris Saint-Joseph, Paris
  - HIA Val-de-Grâce, Paris
  - Hôpital Bichat - Claude - Bernard, Paris
  - Paris - Curie, Paris
  - Pau - CH, Pau
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - CHU, Poitiers
  - Pontoise - CH, Pontoise
  - Quimper - CH, Quimper
  - Reims - CHU, Reims
  - Institut Jean Godinot, Reims
  - Rennes - CHU, Rennes
  - Roubaix - CH, Roubaix
  - Saint-Cloud - Centre René Huguenin, Saint-Cloud
  - Saint Priest en Jarez - ICL, Saint-Priest-en-Jarez
  - Saint Quentin - CH, Saint-Quentin
  - Salon de Provence - CH, Salon-de-Provence
  - Sens - CH, Sens
  - Strasbourg - NHC, Strasbourg
  - Thonon les bains - CH, Thonon-les-Bains
  - Toulon - CHI, Toulon
  - Toulon - HIA, Toulon
  - Toulouse - CHU Larrey, Toulouse
  - Tourcoing - CH, Tourcoing
  - Tours - CHU, Tours
  - Valenciennes - Clinique, Valenciennes
  - Versailles - CH, Versailles
  - CHI de la Haute-Saône - Pneumologie, Vesoul
  - CH de Villefranche - Pneumologie, Villefranche
  - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Souquet PJ, Audigier-Valette C, Molinier O, Cortot A, Margery J, Moreau L, Gervais R, Barlesi F, Pichon E, Zalcman G, Dumont P, Girard N, Poudenx M, Mazieres J, Cadranel J, Debieuvre D, Dauba J, Langlais A, Morin F, Moro-Sibilot D, Westeel V, Perol M. Tailoring maintenance chemotherapy upon response to induction chemotherapy as compared with pemetrexed continuation maintenance in advanced non-squamous NSCLC patients: Results of the IFCT-GFPC-1101 multicenter randomized phase III trial. Lung Cancer. 2022 Feb;164:84-90. doi: 10.1016/j.lungcan.2021.11.014. Epub 2021 Nov 30. PMID 35051725
- See also: IFCT official website — http://www.ifct.fr